CLINICAL TRIAL: NCT00909727
Title: A Phase 3, 2-Part, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Pharmacokinetics, Efficacy and Safety of VX-770 in Subjects Aged 6 to 11 Years With Cystic Fibrosis and the G551D Mutation
Brief Title: Study of Ivacaftor in Cystic Fibrosis Subjects Aged 6 to 11 Years With the G551D Mutation
Acronym: ENVISION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX08-770-103
Record Dates: First submitted 2009-05-26; First posted 2009-05-28 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Cystic Fibrosis
Keywords: Fibrosis; Pancreatic Diseases; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes
MeSH Terms: conditions — Cystic Fibrosis; Fibrosis; Pancreatic Diseases; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Pathologic Processes | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects who received placebo every 12 hours (q12h) for up to 48 weeks.
  Interventions: Drug: Placebo
- 150 mg Ivacaftor q12h (Experimental): Subjects who received 150 mg of ivacaftor q12h for up to 48 weeks.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor — 150-mg tablet given orally q12h for up to 48 weeks
  Other Names: VX-770
  Arms: 150 mg Ivacaftor q12h
Drug: Placebo — Tablet given orally q12h for up to 48 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of ivacaftor in subjects with cystic fibrosis aged 6 to 11 years who have the G551D mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene. Ivacaftor is a potent and selective potentiator of wild-type, G551D, F508del, and R117H forms of human CFTR protein. Potentiators are pharmacological agents that increase the chloride ion transport properties of the channel in the presence of cyclic adenosine monophosphate (AMP)-dependent protein kinase A (PKA) activation.

DETAILED DESCRIPTION:
This is a Phase 3, 2-part, randomized, double-blind, placebo-controlled, parallel group multicenter study of orally administered ivacaftor in subjects with cystic fibrosis (CF) 6 to 11 years of age who have the G551D-CFTR mutation and a forced expiratory volume in 1 second (FEV1) between 90% and 105% predicted (using Knudson standards).

Based on in vitro studies and pharmacologic, pharmacokinetic (PK), and safety profiles, ivacaftor was selected for clinical development as a possible treatment for patients with CF. Patients with the G551D mutation were the targeted population for this study because ivacaftor is a potentiator of the gating effect of the CFTR protein, and the most prevalent mutation with a gating defect in CF is the G551D mutation.

This study was conducted in 2 parts. Part A was conducted to analyze the PK properties of ivacaftor and to determine the most appropriate dose to administer to subjects in Part B of this study. Part B explored the safety and efficacy of ivacaftor over long-term treatment in subjects 6 to 11 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Weighing at least 15 kg
* Confirmed diagnosis of cystic fibrosis (CF) and G551D mutation in at least 1 allele
* Forced expiratory volume in 1 second (FEV1) of 40% to 105% (inclusive) of predicted normal for age, gender, and height (Knudson standards) at Screening
* Able to swallow tablets
* As judged by the investigator, parent or legal guardian and subject must have been able to understand protocol requirements, restrictions, and instructions, and the parent or legal guardian should have been able to ensure that the subject complied with, and was likely to complete, the study as planned
* Parent or legal guardian must have signed the informed consent form and corresponding assent must be obtained from the subject
* Willing to use at least 1 highly effective birth control method during the study
* No clinically significant abnormalities that would have interfered with the study assessments, as judged by the investigator

Exclusion Criteria:

* History of any illness or condition that might confound the results of the study or pose an additional risk in administering study drug to the subject
* Acute respiratory infection, pulmonary exacerbation, or changes in therapy for pulmonary disease within 4 weeks of Day 1 of the study
* Abnormal liver function ≥ 3x the upper limit of normal
* Abnormal renal function at Screening
* History of solid organ or hematological transplantation
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within 30 days prior to Screening
* Use of inhaled hypertonic saline treatment
* Concomitant use of any inhibitors or inducers of cytochrome P450 3A4 (CYP 3A4)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ahrens, MD, Principal Investigator — Roy A. & Lucille A. Carver College of Medicine
Locations (29):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - Emory Cystic Fibrosis Center, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - The Cystic Fibrosis Center of Chicago, Glenview, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Department of Pediatrics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Helen DeVos Children's Hospital Spectrum Health Hospitals, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center Pediatric Pulmonary/ CF, Omaha, Nebraska
  - East Tennessee Children's Hospital Pediatric Pulmonary and Respiratory Care, Knoxville, Tennessee
  - University of Utah Pediatric Pulmonology, Salt Lake City, Utah
  - University of Virginia Pediatric Respiratory Medicine, Charlottesville, Virginia
- Australia (4):
  - The Children's Hospital Westmead, Westmead, New South Wales
  - Royal Children's Hospital Brisbane, Herston, Queensland
  - Royal Children's Hospital Melbourne, Parkville, Victoria
  - Princess Margaret Hospital for Children, Subiaco, Western Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital for Sick Children CF Center, Toronto, Ontario
- Hôpital Robert Debré - Service de gastro-entérologiemucoviscidose et nutrition, Paris, France
- Germany (2):
  - Kinder- und Jugendklinik Universitätsklinikum Erlangen, Erlangen
  - Mukoviszidose-Zentrum am Klinikum der Friedrich-Schiller-Universität Jena, Klinik für Kinder- und Jugendmedizin, Jena
- Ireland (2):
  - Our Lady's Children's Hospital, Dublin
  - The National Children's Hospital, Dublin
- Dept of Gene Therapy, Imperial College London, London, United Kingdom

REFERENCES:
- [Derived] Davies JC, Wainwright CE, Canny GJ, Chilvers MA, Howenstine MS, Munck A, Mainz JG, Rodriguez S, Li H, Yen K, Ordonez CL, Ahrens R; VX08-770-103 (ENVISION) Study Group. Efficacy and safety of ivacaftor in patients aged 6 to 11 years with cystic fibrosis with a G551D mutation. Am J Respir Crit Care Med. 2013 Jun 1;187(11):1219-25. doi: 10.1164/rccm.201301-0153OC. PMID 23590265
- See also: Genetics Home Reference — http://ghr.nlm.nih.gov/
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part A started on 05 August 2009 (signing of first informed consent). Screening evaluations were completed during Day -28 to Day -2. All subjects completing Part A were offered the opportunity to participate in Part B, which started on 12 March 2010. Screening evaluations were completed during Day -35 to Day -15 before the first dose of study drug.
Pre-assignment Details: Nine subjects were dosed and included in Part A. In Part B, 52 subjects were enrolled and all were randomized to ivacaftor (26 subjects) or placebo (26 subjects). A 2-week run-in period was included to establish the baseline assessments on Day 1 after ensuring that subjects were properly taking their cystic fibrosis (CF) medication regimens.
Groups:
- Placebo: Oral tablet every 12 hours (q12h) for up to 48 weeks
- 150 mg Ivacaftor q12h: Oral tablet of 150 mg of ivacaftor q12h for up to 48 weeks
Period: Overall Study
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Started | 26 (All subjects who received at least 1 dose of study drug (placebo)) | 26 (All subjects who received at least 1 dose of study drug (ivacaftor))
Completed Treatment Period, Week 24 | 23 | 26
Completed | 22 (Completed Treatment and Extension Periods (through Week 48)) | 26 (Completed Treatment and Extension Periods (through Week 48))
Not Completed | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Wrong Genotype | 1 | 0
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Prohibited Medication | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 150 mg Ivacaftor q12h | Total
Number analyzed (Participants) | 26 | 26 | 52
Age Continuous [Mean (Standard Deviation); unit: years] | 8.9 (1.86) | 8.9 (2.00) | 8.9 (1.91)
Age, Customized [Number; unit: participants]
  6 to 8 Years | 13 | 12 | 25
  9 to 11 Years | 12 | 11 | 23
  > 11 Years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 16 | 9 | 25
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23 | 22 | 45
  Other | 1 | 2 | 3
  Not Allowed to Ask Per Local Regulations | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 24 | 23 | 47
  Not Allowed to Ask Per Local Regulations | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  North America | 15 | 12 | 27
  Europe | 5 | 6 | 11
  Australia | 6 | 8 | 14
Weight [Mean (Standard Deviation); unit: kilograms] | 30.0 (7.16) | 31.8 (9.95) | 30.9 (8.63)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 16.8 (1.75) | 17.1 (2.61) | 17.0 (2.21)
Sweat Chloride [Mean (Standard Deviation); unit: millimoles per liter] | 104.8 (8.87) | 104.3 (14.54) | 104.6 (11.92)
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Number; unit: participants] — Percent predicted for age, gender, and height
  participants
    < 70% | 8 | 4 | 12
    ≥ 70% to ≤ 90% | 6 | 12 | 18
    > 90% | 12 | 10 | 22
Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: percentage] — Percent predicted for age, gender, and height
  percentage | 83.7 (20.37) | 84.7 (15.83) | 84.2 (18.07)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 24
Description: Spirometry (as measured by FEV1) is a standardized assessment to evaluate lung function that is the most widely used endpoint in cystic fibrosis studies.
Time Frame: baseline through 24 weeks
Population: All randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo)and had available assessments during the time frame.
Measure: Least Squares Mean (Standard Error); unit: percent of predicted volume (L)
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 25 | 26
percent of predicted volume (L) | 0.1 (2.1) | 12.6 (2.1)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; The primary analysis for the primary efficacy variable was based on a Mixed-Effects Model for Repeated Measures (MMRM). The model included absolute change from baseline in percent predicted forced expiratory volume in 1 second (FEV1) as the dependent variable, treatment (ivacaftor versus placebo) and visit (Day 15, Week 8, Week 16, and Week 24) as fixed effects, and subject as a random effect, with adjustment for the continuous baseline value of percent predicted FEV1; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The primary endpoint and key secondary endpoints were tested in sequence. test 1: primary (α=0.05); test 2: using Hochberg's step-up procedure on weight (Wk 24) and sweat chloride (Wk 24)(α=0.05); test 3: CFQ-R respiratory domain score (Wk 24); Denominator degrees of freedom were estimated using the Kenward-Roger approximation. No imputation of missing data was done; Mean Difference (Final Values) = 12.5, 95% CI 2-sided [6.6 to 18.3], Standard Error of Mean 2.9

2. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 48
Description: as for outcome 1
Time Frame: baseline through 48 weeks
Population: All randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo) and had available assessments during the time frame.
Measure: Least Squares Mean (Standard Error); unit: percent of predicted volume (L)
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 25 | 26
percent of predicted volume (L) | 0.7 (2.0) | 10.7 (1.9)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint, a Mixed-Effects Model for Repeated Measures (MMRM). Estimates were obtained from MMRM with dependent variable absolute change from baseline, fixed effects for categorical visit & treatment group, & adjustment for the continuous baseline value of percent predicted FEV1, using unstructured covariance matrix; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — There was no adjustment for multiple comparisons; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.0, 95% CI 2-sided [4.5 to 15.5], Standard Error of Mean 2.7

3. Secondary Outcome: Absolute Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Through Week 24 and Week 48 (Respiratory Domain Score, Children)
Description: The CFQ-R is a health-related quality of life measure for subjects with cystic fibrosis. Each domain is scored from 0 (worst) to 100 (best). A difference of at least 4 points in the respiratory domain score of the CFQ-R is considered a minimal clinically important difference (MCID).
Time Frame: baseline through 24 weeks and 48 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 25 | 26
score on a scale
  Change from Baseline Through Week 24 | 0.3 (2.6) | 6.3 (2.5)
  Change from Baseline Through Week 48 | 1.0 (2.3) | 6.1 (2.2)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 24: Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint, a Mixed-Effects Model for Repeated Measures (MMRM), with the addition of the baseline domain score as a covariate; Test type: Superiority or Other; p = 0.1092, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.1, 95% CI 2-sided [-1.4 to 13.5], Standard Error of Mean 3.7
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 48: Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint, a Mixed-Effects Model for Repeated Measures (MMRM), with the addition of the baseline domain score as a covariate; Test type: Superiority or Other; p = 0.1354, Mixed Models Analysis — There was no adjustment for multiple comparisons; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [-1.6 to 11.8], Standard Error of Mean 3.3

4. Secondary Outcome: Absolute Change From Baseline in Sweat Chloride Concentration Through Week 24 and Week 48
Description: The sweat chloride (quantitative pilocarpine iontophoresis) test is a standard diagnostic tool for cystic fibrosis (CF), serving as an indicator of cystic fibrosis transmembrane conductance regulator (CFTR) activity.
Time Frame: baseline through 24 weeks and 48 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 23 | 23
millimoles per liter
  Change from Baseline Through Week 24 | -1.2 (2.6) | -55.5 (2.6)
  Change from Baseline Through Week 48 | -2.6 (2.6) | -56.0 (2.5)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 24: Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous baseline value for sweat chloride and percent predicted forced expiratory volume in 1 second (FEV1), using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -54.3, 95% CI 2-sided [-61.8 to -46.8], Standard Error of Mean 3.7
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; Through Week 48: Analysis for this variable was similar to that of the primary analysis of the primary efficacy endpoint. Estimates were from Mixed-Effects Model for Repeated Measures (MMRM) with dependent variable absolute change from baseline, fixed effects for categorical visit and treatment group, and adjustment for continuous baseline value for sweat chloride and percent predicted forced expiratory volume in 1 second (FEV1), using unstructured covariance matrix; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — There was no adjustment for multiple comparisons; Mean Difference (Final Values) = -53.5, 95% CI 2-sided [-60.9 to -46.0], Standard Error of Mean 3.7

5. Secondary Outcome: Absolute Change From Baseline in Weight at Week 24 and Week 48
Description: As malnutrition is common in patients with cystic fibrosis (CF) because of increased energy expenditures due to lung disease and fat malabsorption, body weight is an important clinical measure of nutritional status.
Time Frame: baseline to 24 weeks and 48 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Number analyzed (Participants) | 26 | 26
kilograms
  At Week 24 | 1.8 (0.4) | 3.7 (0.4)
  At Week 48 | 3.1 (0.5) | 5.9 (0.5)
Statistical Analysis 1: Comparison: Placebo vs 150 mg Ivacaftor q12h; At Week 24: Analysis for this variable was based on a Linear Mixed Effect (LME) model with dependent variable weight; treatment as a fixed effect; and intercept, visit, and treatment by visit interaction as random effects, with adjustment for baseline percent predicted forced expiratory volume in 1 second (FEV1) severity; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [0.9 to 2.9], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo vs 150 mg Ivacaftor q12h; At Week 48: Analysis for this variable was based on a Linear Mixed Effect (LME) model with random intercept and random slope, treatment as a fixed effect, and visit (days on study) and treatment by visit interaction as random effects, with adjustment for categorical baseline percent predicted forced expiratory volume in 1 second (FEV1) severity; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — P-value is for the treatment effect at Week 48 (obtained as a linear contrast of treatment at Day 336). There was no adjustment for multiple comparisons; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [1.3 to 4.2], Standard Error of Mean 0.7

ADVERSE EVENTS:
Time Frame: For enrolled subjects, adverse events (AEs) were collected through the Follow-up visit in each study part. For subjects who completed 48 weeks of treatment and enrolled in the open-label extension study, AEs were only collected through the Week 48 visit.
Arm/Group | Placebo | 150 mg Ivacaftor q12h
Serious Adverse Events (participants affected / at risk) | 6/26 | 5/26
Other Adverse Events (participants affected / at risk) | 25/26 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | 150 mg Ivacaftor q12h (N=26)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 3 (3) | 2 (2) — CF exacerbations were coded as "cystic fibrosis lung."
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | 150 mg Ivacaftor q12h (N=26)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (40) | 13 (21)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (9) | 7 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 5 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (9)
Bronchitis (Infections and infestations) | 2 (2) | 3 (4)
Otitis media (Infections and infestations) | 1 (2) | 4 (7)
Sinusitis (Infections and infestations) | 3 (4) | 2 (3)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 6 (9)
Vomiting (Gastrointestinal disorders) | 7 (11) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (6) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 3 (3)
Bacteria sputum identified (Investigations) | 3 (3) | 2 (2)
Pulmonary function test decreased (Investigations) | 3 (4) | 2 (2)
Eosinophil count increased (Investigations) | 1 (1) | 3 (5)
Culture throat positive (Investigations) | 1 (1) | 2 (2)
Breath sounds abnormal (Investigations) | 2 (3) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3)
White blood cell count decreased (Investigations) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 7 (16) | 6 (6)
Fatigue (General disorders) | 2 (2) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 2 (3) | 1 (2)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 6 (8) | 7 (9) — CF exacerbations were coded as "cystic fibrosis lung."
Headache (Nervous system disorders) | 4 (8) | 7 (15)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days